CLINICAL TRIAL: NCT06950476
Title: Assisted Reproductive Technology Cycle Outcomes When Only 1 to 3 Oocytes Are Retrieved: a Retrospective Analysis of 3,671 Cycles in Poor Responders From a Large Volume Single Center
Brief Title: ART Cycle Outcomes When Only 1 to 3 Oocytes Are Retrieved
Acronym: POR
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: POOR RESPONDERS
Record Dates: First submitted 2025-04-28; First posted 2025-04-30 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Infertility Assisted Reproductive Technology; Oocyte Retrieval
MeSH Terms: interventions — Oocyte Retrieval

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Oocyte Retrieval — Oocyte retrieval is performed at the end of ovarian stimulation (OS) to collect oocytes for use in IVF or ICSI cycles.

SUMMARY:
This is a monocentric retrospective observational study. The study focuses on the women who underwent Assisted Reproductive Technology (ART) cycles with poor ovarian response (POR), defined as <4 oocytes retrieved.

The objectives of the study are as follows:

* Evaluate clinical pregnancy rate (CPR) and cumulative live birth rate (CLBR) in women with poor ovarian response.
* Evaluate abortion rate in women with poor ovarian response.
* Evaluate the influence of patient characteristics (age, Anti-Müllerian hormone [AMH] levels, Antral Follicle Count [AFC], Follicle Stimulating Hormone [FSH], Body Mass Index [BMI]) on women with poor ovarian response.

To address the study objectives, data will be collected using a specific internal web-based database. All oocyte retrieval procedures performed at the Humanitas Fertility Center from January 2010 to December 2023 will be included in the evaluation. Outcomes will be expressed in terms of CLBR, CPR and Abortion Rate.

ELIGIBILITY:
Inclusion Criteria:

* The study database will include all women who underwent IVF treatment between 2010 and 2023 and were classified as poor ovarian responders, defined as those who retrieved fewer than 4 oocytes following controlled ovarian stimulation.

Exclusion Criteria:

* The study database will exclude women who underwent IVF treatment and retrieved more than 3 oocytes following controlled ovarian stimulation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study sample will include all patients registered in the Humanitas Fertility Center database between January 2010 and December 2023, matching the inclusion and exclusion criteria cited above.
Sampling Method: Probability Sample
Enrollment: 3761 (Actual)
Dates: Start 2010-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Clinical Pregnancy Rate (CPR) | January 2010 - December 2023
  This study aims to evaluate the ART outcomes in women classified as poor ovarian responders (POR), focusing on clinical pregnancy rate.
  The CPR is defined as the number of clinical pregnancies expressed per 100 initiated cycles.
Cumulative Live Birth Rate (CLBR) | January 2010 - December 2023
  This study aims to evaluate the ART outcomes in women classified as poor ovarian responders (POR), focusing on cumulative live birth rates The CLBR is defined as the likelihood of achieving at least one live birth over a series of treatment cycles, including both fresh and frozen embryo transfers, originating from a single ovarian stimulation.
Abortion Rate | January 2010 - December 2023
  This study aims to evaluate the ART outcomes in women classified as poor ovarian responders (POR), focusing on abortion rates.
  Abortion rate is defined as the presence of an empty gestational sac or a gestational sac containing an embryo or fetus without fetal cardiac activity, occurring within the first 12 6/7 weeks of gestation.